CLINICAL TRIAL: NCT00040417
Title: Allo SCT From HLA Haploidentical Related Donors Using Sub-Myeloablative Conditioning For Patients With High Risk Hemoglobinopathies: Hemo SS, Hemo SC, Hemo SB0/+ Thalassemia, Homozygous B0/+ Thalassemia or Severe B0/+ Thalassemia Variants
Brief Title: Bone Marrow Transplant From Donor Using Less Toxic Conditioning for Patient With High Risk Hemoglobinopathies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to accrue patients
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H8750; Smallo
Record Dates: First submitted 2002-06-26; First posted 2002-06-27 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Anemia; Hemoglobinopathy; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; Thalassemia | interventions — fludarabine; Whole-Body Irradiation; Tacrolimus; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: FLUDARABINE
Drug: CAMPATH-IH
Procedure: Total Body Irradiation
Drug: FK506
Drug: G-SCF (Granulocyte-colony stimulating factor)

SUMMARY:
The major goal of this study is to determine the risks and benefits of stem cell transplants in combination with a newer, less toxic conditioning chemotherapy treatment in patients with severe sickle cell disease (SCD) or sickle hemoglobin variants (hemoglobin SC or hemoglobin SB0/+), or homozygous b0/+ thalassemia or severe B0/+ thalassemia variants. Participation in this project will be for one year, with follow up evaluations done every 6 months thereafter for 10 years or until participants are 18 years old.

DETAILED DESCRIPTION:
To do the stem cell transplant, we must first kill most of the cells in the bone marrow that make the sickle hemoglobin or abnormal blood cells of severe beta thalassemia. We will do this by using a single dose of body irradiation and two drugs called Fludarabine and Campath-IH.

The treatment schedule is as follows:

Day - 6: Total body irradiation Day - 5: Fludarabine and Campath 1H Day - 4: Fludarabine and Campath 1H Day - 3: Fludarabine and Campath 1H Day - 2: Fludarabine and Campath 1H Day - 1: REST Day 0: Stem Cell Transplant (infusion)

After the drug treatment, participants will be given healthy stem cells from a related donor that partially matches their HLA (immune) type, most likely from a parent or sibling. This is known as the stem cell transplant.

The healthy stem cells will be put into a blood vein in the same way that transfusions are given. The cells then travel to the right places in the body, where they should grow and make new blood cells that do not sickle.

ELIGIBILITY:
Inclusion:

* Patients with a haploidentical related HLA donor and hemoglobin SS, hemoglobin SC, or hemoglobin Sb0/+ thalassemia and at least one of the following conditions:

  1. previous central nervous system vaso-occlusive episode with or without residual neurologic findings;
  2. frequent painful vaso-occlusive episodes which significantly interfere with normal life activities and which necessitate chronic transfusion therapy;
  3. recurrent SCD chest syndrome events, which necessitate chronic transfusion therapy;
  4. severe anemia, which prevents acceptable quality of life and necessitates chronic transfusion therapy.
* Patients with a haploidentical related HLA donor and homozygous b0/+ thalassemia or severe variants of b0/+ thalassemia and require chronic transfusion therapy.
* Women of childbearing potential must have a negative pregnancy test.
* Between the ages of birth and 65 years.

Exclusion:

* HLA identical or 5/6 HLA matched sibling donor
* Biopsy proven chronic active hepatitis or portal fibrosis.
* SCD chronic lung disease > stage 3 Severe renal dysfunction defined as creatinine clearance <40 ml/min/1.73 M2.
* Severe cardiac dysfunction defined as shortening fraction <25%.
* HIV infection.
* Unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate Stem Cell Transplant.
* Patient or guardian(s) unable to understand the nature and risks inherent in the stem cell transplant process.
* Pregnant or lactating females and those unwilling to use acceptable contraception.

Ages: 1 Day to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2000-08; Primary Completion 2003-11-21 (Actual); Study Completion 2003-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K. Brenner, MD, FRCP, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas